CLINICAL TRIAL: NCT06419322
Title: A Monocentric, Prospective and Longitudinal Study Investigating the Acceptability, Feasibility, Safety and Efficacy of an Optimized Rehabilitation Program for Treated Patients With SMA Compared to the Current Rehabilitation Program in United Kingdom: ACE SMA.
Brief Title: Acceptability, Feasibility, Safety and Efficacy of a Optimized Rehabilitation Program for Treated Patients With Spinal Muscular Atrophy (SMA).
Acronym: ACE SMA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford Brookes University (Other); Oxford University Hospitals NHS Trust (Other); ACE SMA Charity (Unknown); Roche Products Limited (Unknown); Scholar Rock, Inc. (Industry); Biohaven Therapeutics Ltd. (Industry); Rally Round Rupert Charity (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACE SMA; PID17165 (Other: University Oxford Hospitals NHS Foundation Trust)
Record Dates: First submitted 2024-05-02; First posted 2024-05-17 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-05

CONDITIONS: Spinal Muscular Atrophy
Keywords: physiotherapy; rehabilitation; SMA; acceptability; feasibility; United Kingdom; physical therapy; prospective; Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Intervention Model Description: All participants will receive the optimized rehabilitation program (intervention). An external control group will be used to determine the potential efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated cohort (Other)
  Interventions: Other: Optimized rehabilitation program

INTERVENTIONS:
Other: Optimized rehabilitation program — Consisting of: goal-oriented rehabilitation, hands on physiotherapy sessions and home use of SMA approved rehabilitation device.

SUMMARY:
The goal of this study is to investigate the acceptability, feasibility, safety and efficacy of an optimized rehabilitation program for treated patients with spinal muscular atrophy (SMA) compared to the current rehabilitation program in the United Kingdom. The aim is to provide patients with more hands on physiotherapy and access to rehabilitation devices at home to support parents currently providing rehabilitation on their own.

DETAILED DESCRIPTION:
The main study objective is to investigate whether an optimized rehabilitation program would be accepted and is feasible within the SMA patient community.

The optimized program will comprise of goal orientated rehabilitation with more frequent hands on physiotherapy (every 2 weeks) as well as a SMA approved rehabilitation device used at home on a weekly basis, to provide the most appropriate therapy for each individual patient. All study participants will receive the optimized rehabilitation program over 12 months. An external control group will be used to determine the potential efficacy.

Research study visits will take place at baseline, month 6 and month 12. At these visits a general physical exam will be undertaken alongside collecting the participant and carer perception, satisfaction and compliancy of the rehabilitation program. Motor function assessments according to age and ambulatory status will be assessed to help evaluate potential therapeutic benefits.

ELIGIBILITY:
Patient participant Eligibility Criteria:

Inclusion Criteria:

* Genetically confirmed SMA considered as a non-sitter, sitter or walker
* Post-symptomatically treated and on stable dose for 12 months with any disease-modifying market-approved drug
* Patients from 1-10 years of age at baseline
* Parent(s)/legal guardian(s) of patients less than 16 years of age must provide written informed consent prior to the patient's participation in the study
* Willing and able to comply with all protocol requirements and procedures.

Exclusion Criteria:

The participant may not enter the trial if ANY of the following apply:

* Any acute or chronic condition which, as assessed by the investigator, significantly interferes with the rehabilitation of the patient
* Need of diurnal and/or invasive ventilation, naps excluded
* Currently enrolled in a treatment study; or treatment with an experimental therapy
* Any surgical and/or medical intervention, according to the investigator, 3 months before baseline and/or during the study participation.

Carer (considered as participant) Eligibility Criteria:

Inclusion Criteria:

* Willing and able to comply with all protocol requirements and procedures
* Carer's child has been included in study.

Exclusion Criteria:

• No exclusion criteria.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability of an optimized rehabilitation program. Measured as number of eligible patients who accepted to participate in the study compared to the number of eligible patients who have refused to participate. Endpoint: 70% of acceptability. | Baseline visit
  Number of eligible patients who accepted to participate in the study compared to the number of eligible patients who have refused to participate.
Feasibility of an optimized rehabilitation program. Measured as the number of patients who complete the study compared to the number of included patients. Endpoint: 60% of feasibility. | Month 12 (end of study)
  Number of patients who complete the study compared to the number of included patients.

SECONDARY OUTCOMES:
Safety of an optimized rehabilitation program. Measured as the number of serious adverse events (SAE) compared to the year before the baseline. | From baseline to month 12 (end of study)
  Number of Serious Adverse Events (SAEs).
Carer perception and satification measured through the Clinical Global Impression scale - Improvement (CGI I). Comparison of CGI-S score with CGI-I score of the treated group. | Month 6 and Month 12 (end of study).
  Potential effects of the optimized rehabilitation program on patients experience.
Carer perception and satification measured through the Clinical Global Impression scale - Severity (CGI-S). Comparison of CGI-S score with CGI-I score of the treated group. | Baseline visit: CGI-S.
  Potential effects of the optimized rehabilitation program on patients experience.

OTHER OUTCOMES:
The Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND): maximum score is 64 points. Measuring a change in functional total score between the treated study cohort and a control dataset. | Baseline, Month 6, Month 12 (end of study).
  Evaluation potential therapeutic benefits through assessment of motor functional scales.
The Hammersmith Infant Neurological Examination section 2 (HINE-2): maximum score is 26 points. Measuring a change in functional total score between the treated study cohort and a control dataset. | Baseline, Month 6, Month 12 (end of study).
  Evaluation potential therapeutic benefits through assessment of motor functional scales.
Revised Hammersmith Scale (RHS). The maximum score for RHS is 69 points. Measuring a change in functional total score between the treated study cohort and a control dataset. | Baseline, Month 6, Month 12 (end of study).
  Evaluation potential therapeutic benefits through assessment of motor functional scales.
Hammersmith Functional Motor Scale Expanded (HFMSE) combined assessment. The maximum score is 66 points. Measuring a change in functional total score between the treated study cohort and a control dataset. | Baseline, Month 6, Month 12 (end of study).
  Evaluation potential therapeutic benefits through assessment of motor functional scales.
World Health organization (WHO) developmental milestones: the final result is the highest achievable motor milestone. Measuring a change in functional total score between the treated study cohort and a control dataset. | Baseline, Month 6, Month 12 (end of study).
  Evaluation potential therapeutic benefits through assessment of motor functional scales.
Revised upper limb module (RULM): from 30 months of age: maximum score is 37 points. Measuring a change in functional total score between the treated study cohort and a control dataset. | Baseline, Month 6, Month 12 (end of study).
  Evaluation potential therapeutic benefits through assessment of motor functional scales.
6 Minute Walk test (6MWT): from 4 years of age. Measuring a change in functional total score between the treated study cohort and a control dataset. | Baseline, Month 6, Month 12 (end of study).
  Evaluation potential therapeutic benefits through assessment of motor functional scales.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Lilien, Principal Investigator — University of Oxford, Department of Paediatrics
Locations (1):
- Oxford Brookes University, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No